CLINICAL TRIAL: NCT06625463
Title: Development and Implementation Model of Home Based Cardiac Rehabilitation With Family Empowerment Approach in Patient With ACS (HBCR in ACS)
Acronym: HBCR in ACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Eva Marti,Ns.,M.Kep, Mrs.Eva Marti.,S.Kep.,Ns.,M.Kep, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Eva marti 1
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Home Based Rehabilitation; Acute Coronary Syndromes
Keywords: home based cardiac rehabilitation; FCEM; acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking could not be done for researchers and research subjects, but was done for enumerators and assessors of research outcomes. During the data collection and measurement process, enumerators and cardiologists did not know the allocation of research subjects. Likewise, the statistician who will process the data does not know the allocation for each research data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Experimental arm receive 12 week home based cardiac rehabilitation include physical exercise, dietary management, smoking cessation and stress management
  Interventions: Behavioral: Home based cardiac rehabilitation
- control arm (No Intervention): Control arm receive usually care

INTERVENTIONS:
Behavioral: Home based cardiac rehabilitation — 12 week home based cardiac rehabilitation include Physical exercise, dietary management, smoking cessation and stress management
  Arms: Experimental arm

SUMMARY:
The aim of this clinical trial is to determine whether home-based cardiac rehabilitation with a family empowerment approach can help acute coronary syndrome patients recover. The main questions to be answered are:

- Does home-based cardiac rehabilitation with a family approach effective in patients with acute coronary syndrome to improve health-related quality of life and peak Vo2? Researchers will compare with usual care to see if home-based cardiac rehabilitation with a family approach is more effective for improving health-related quality of life and peak Vo2 in ACS patients.

Patient inclusion criteria

1. Patients with acute coronary syndrome who had undergone hospitalization, with a minimum home care time of 3 months and a maximum of 1 year, calculated from the day of discharge from the hospital until the time of the interview.
2. Aged 18-65 years old, participants were selected with age variations representing young adults, adults and the elderly.
3. Patients with first experience of SCA, participants were selected whether they had undergone PCI or not.
4. Patients living with family and family involved in the patient care process.
5. Physical condition allows for interviews. physical condition is evidenced by examination of stable vital signs (diastolic BP

   >90, systolic <150 mmhg; N: 60-100x/min; S: 36-380c, no pain). Psychological condition does not show symptoms of depression as measured by the Patient Health Questionnaire-9 instrument.
6. Willing to participate in the study.

Participants will:

For 12 weeks

1. Perform walking exercises as prescribed
2. Implement diets and stress management according to the module
3. Quit smoking
4. Medication compliance
5. visit the clinic to see a cardiologist, undergo a 6-minute walk test

DETAILED DESCRIPTION:
How to enroll patients as research subjects Inpatients

1. The research team determines SKA patients who fit the study criteria
2. The room nurse helps explain to the patient to be involved in the study, explaining the purpose, benefits, procedures of the study and possible risks
3. The room nurse will ask the patients willingness to be involved in the study.
4. The patient signs the Informed consent
5. The nurse explains the interventions that will be provided after informed consent during the first hospital visit (details of the interventions are in the next section).
6. The nurse will give the prospective research subject identification card to the family and convey it to the outpatient clinic nurse.

Outpatients

1. The research team draws data from medical records and determines appropriate outpatients. With criteria
2. The research team gave a list of patients who could be used as research subjects to the outpatient nurse on duty
3. The nurse will help explain to the patient to be involved in the study, explaining the purpose, benefits, procedures of the study and the risks that may occur
4. The room nurse will ask for the patients willingness to be involved in the study.
5. The patient signs the Informed consent

Intervention HBCR with FCEM approach

1. Baseline measurement and entry test stage
2. At this stage, peak VO2 measurement is taken, measured based on 6MWT travel time. The results of the 6-minute walk test will be used to determine the intensity of home exercise to be performed. The research subjects will undergo ECG examination before and after the 6MWT to ensure the following
3. Patients and families will receive the HBCR module, which consists of a guidebook and educational video at the beginning of the counselling education session.
4. Patients and families receive a video by a cardiologist explaining. disease and treatment, a video by a psychologist on stress management, a dietician on food management, aiming to maintain weight and blood sugar levels and a video on smoking cessation guidance by a smoking counsellor.
5. Family-centered empowerment education stage

   * Explain the threat of ACS, signs and symptoms, clinical manifestations, complications, treatment and follow-up care, risk factor control, and the role of the family in home-based cardiac rehabilitation (all families in the intervention group).
   * Patients and families are guided by 1 facilitator. In the group, an intervention to increase self-efficacy was conducted by exploring problems that might arise in advanced care, and then exploring joint solutions to these problems.
   * Interventions to improve self-esteem and family participation were conducted. Family members were educated based on the distributed module on controlling the risk of SCA patients in cardiac rehabilitation, practiced how to accompany and monitor patients in cardiac rehabilitation Given positive reinforcement and feedback. The group also ensures the family's correct understanding in managing cardiac rehabilitation at home through a question and answer session.
   * The facilitator evaluates the process and results of the stages that have been carried out to family members.
6. 12 weeks Home-based Cardiac Rehabilitation

   1. The hbcr session is 12 weeks, the patient will be seen by the cardiologist at weeks 1, 6, 12. During the 12-week intervention process, the cardiologist in charge of the patient is the same cardiologist who performed the risk assessment examination on the patient, determining the activity based on the first 6MWT test performed by the patient. During the intervention process, the facilitating nurse will report to the cardiologist in charge if there is any deterioration in the patiens condition, in terms of vital signs and activities.
   2. Smoking, diet and stress management counseling was conducted at the beginning of the session, and follow-up by the nurse every 2 weeks in month 1, and every 4 weeks in the following month (in the form of follow-up per video call/home visit). Visit every 4 weeks to the cardiologist
   3. Physical exercise is done 3 times a week, 1 session of 30-40 minutes. Patients can choose from jogging, cycling, weight lifting or aerobic exercise. Each exercise session consists of 5 minutes of warm-up, 30 minutes of core exercise and 5 minutes of cool-down. Patients and families are given a video on the direction of the physical exercise to be performed. Each exercise is accompanied by the family, to monitor the patients HR, complaints during the exercise session.
   4. The family reports HR and complaints during exercise, immediately after the exercise is performed
   5. The family reports daily diet, exercise frequency, complaints on the form provided.

During the intervention period, the family reported daily diets, medication adherence and exercise activities as well as HR during exercise through a daily google form that would be monitored by the facilitating nurse.

The control group will receive education on the components of medication adherence, exercise, smoking behaviour, diet, and stress management for 1 session.

Forms of protection for patients and families:

1. Informed consent is given in detail, clearly and easily understood by patients and families.
2. Confidentiality of patient and family data
3. Patients and families have the right to resign during the research process.
4. Families are trained and enabled to provide home-based cardiac rehabilitation assistance to patients before the intervention is carried out.
5. The activity plan given to patients is in accordance with their abilities, as measured by the 6MWT test. Patients who participated were patients with mild and moderate categories.
6. There is one cardiologist who is in charge of the intervention and a nurse facilitator who will conduct daily monitoring through g forms, monitoring every two weeks through video calls or home visits. Nurse facilitators have previously been trained.
7. There is a prepared flow in case of an emergency situation, by coordinating with the nearest health care centre to the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute coronary syndrome who have undergone hospitalization, with a minimum home care time of 3 months and a maximum of 1 year, calculated from the day of discharge from the hospital until the time of interview.
2. Aged 18-65 years, participants were selected with age variations representing young adults, adults and the elderly.
3. Patients with first experience of SCA, participants were selected whether they had undergone PCI or not.
4. Patients living with family and family involved in the patient care process.
5. Physical condition allows for interviews. physical condition is evidenced by examination of stable vital signs (diastolic BP

   >90, systolic <150 mmhg; N: 60-100x/min; S: 36-380c, no pain). Psychological condition does not show symptoms of depression as measured by the Patient Health Questionnaire-9 instrument.
6. Willing to participate in the study.

Exclusion Criteria:

* Patients with comorbidities that require routine medication such as Diabetes Mellitus, hypertension, renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
health related quality of life | From enrollment to the end of treatment at 12 weeks
  Individuals perception of their level of health, current condition which includes physical, psychological and social dimensions, will be measured with MacNew Heart questionnaire. scored from 1 (low HRQOL) to 7 (high HRQOL). The maximum possible score in any domain is 7
peak Vo2 | From enrollment to the end of treatment at 12 weeks
  peak vo2 achieved based on 6minute walk test, in ml/kg/min

CONTACTS AND LOCATIONS:
Overall Officials: Anggoro Budi Hartopo, PhD, Study Director — Gadjah Mada University
Locations (2):
- Indonesia (2):
  - Gadjah Mada University, Sleman, Special Region of Yogyakarta
  - Rsup Dr Sardjito, Yogyakarta, Special Region of Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basuki N, El-Ansary D, Hofer S, Dwiputra B, Nualnim N. The Validity and Reliability of the MacNew Heart Disease Health Related Quality of Life Questionnaire: The Indonesian Version. Acta Med Indones. 2021 Jul;53(3):276-281. PMID 34611066
- [Background] Arena R, Myers J, Williams MA, Gulati M, Kligfield P, Balady GJ, Collins E, Fletcher G; American Heart Association Committee on Exercise, Rehabilitation, and Prevention of the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing. Assessment of functional capacity in clinical and research settings: a scientific statement from the American Heart Association Committee on Exercise, Rehabilitation, and Prevention of the Council on Clinical Cardiology and the Council on Cardiovascular Nursing. Circulation. 2007 Jul 17;116(3):329-43. doi: 10.1161/CIRCULATIONAHA.106.184461. Epub 2007 Jun 18. No abstract available. PMID 17576872
- [Background] Alhani F, Asghari-Jafarabadi M, Norouzadeh R, Rahimi-Bashar F, Vahedian-Azimi A, Jamialahmadi T, Sahebkar A. The effect of family-centered empowerment model on the quality of life of adults with chronic diseases: An updated systematic review and meta-analysis. J Affect Disord. 2022 Nov 1;316:140-147. doi: 10.1016/j.jad.2022.07.066. Epub 2022 Aug 11. PMID 35964767